CLINICAL TRIAL: NCT03792347
Title: A Phase Ib Study of Pre-Operative Pembrolizumab + Chemoradiation in Patients With Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Preoperative Anti-PD-1 Antibody Combined With Chemoradiotherapy for Locally Advanced Squamous Cell Carcinoma of Esophagus
Acronym: PALACE-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hecheng Li M.D., Ph.D (Other)
Responsible Party: Sponsor-Investigator, Hecheng Li M.D., Ph.D, Professor, Ruijin Hospital
Organization: Ruijin Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTS-007
Record Dates: First submitted 2018-12-28; First posted 2019-01-03 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: esophageal squamous cell carcinoma; neoadjuvant chemoradiotherapy; pembrolizumab; immune therapy; checkpoint inhibitor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Participants will receive carboplatin (AUC=2) IV and paclitaxel (50mg/m²) IV on day 1,8,15,22,29. And radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week. Participants will also receive pembrolizumab (2mg/kg) IV on days 1 and 22. Surgery will be performed within 6 weeks after completion of preoperative therapy described above
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Arm 1:preoperative pembrolizumab with chemoradiotherapy group Participants will receive carboplatin (AUC=2) IV and paclitaxel (50mg/m²) IV on day 1,8,15,22,29. And radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week. Participants will also receive pembrolizumab (2mg/kg) IV on days 1 and 22. Surgery will be performed within 6 weeks after completion of preoperative therapy described above.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Arm1：Pre-operative Pembrolizumab+chemoradiotherapy
  Other Names: Keytruda

SUMMARY:
This study will evaluate the safety and feasibility of preoperative immune checkpoint therapy with concurrent chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma. And this study will provide valuable information for further clinical trials of preoperative pembrolizumab and other immune checkpoint therapy in esophageal cancer treatment.

DETAILED DESCRIPTION:
Esophageal cancer ranks the eighth most common cancer (the fifth most common cancer in China), while ESCC is the most common subtype in Asia (more than 90 % in china). Radical resection is thought to be the mainstay of esophageal cancer treatment and preoperative CRT is well applied in treating locally advanced esophageal cancer. In a multicohort, phase IB study, pembrolizumab was used in 23 unresectable esophageal cancer patients. In this clinical trial, the incidence of grade 3 treatment-related adverse events was 39 % without the appearance of grade 4 and higher-grade adverse event, while the overall response rate reached 30 %. The safety of immune checkpoint therapy for unresected esophageal cancers using nivolumab, a different PD-1 monoclonal antibody, has also been confirmed by high quality clinical trials.

This study will evaluate the safety and feasibility of preoperative immune checkpoint therapy using pembrolizumab with concurrent chemoradiotherapy in patients with locally advanced esophageal squamous cell carcinoma. And this study will provide valuable information for further clinical trials of preoperative pembrolizumab and other immune checkpoint therapy in esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* A patient will be eligible for inclusion in this study only if ALL of the following criteria apply:

  1. Histologically confirmed cT2-T4a,N0-N+,M0 resectable esophageal squamous cell carcinoma
  2. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
  3. Patients approve and sign the informed consent

Exclusion Criteria:

* 1. Patients with active autoimmune disease or history of autoimmune disease 2. Patients who have a condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications 3. Subjects with a history of symptomatic interstitial lung disease 4. History of allergy to study drug components 5. Women must not be pregnant or breast-feeding 6. Men with female partners (WOCBP) that are not willing to use contraception 7. Patient has received prior chemotherapy, radiotherapy, target therapy and immune therapy for this malignancy or for any other past malignancy 8. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hecheng Li, MD PHD, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li C, Zhao S, Zheng Y, Han Y, Chen X, Cheng Z, Wu Y, Feng X, Qi W, Chen K, Xiang J, Li J, Lerut T, Li H. Preoperative pembrolizumab combined with chemoradiotherapy for oesophageal squamous cell carcinoma (PALACE-1). Eur J Cancer. 2021 Feb;144:232-241. doi: 10.1016/j.ejca.2020.11.039. Epub 2020 Dec 26. PMID 33373868

RESULTS

PARTICIPANT FLOW:
Groups:
- Preoperative Pembrolizumab With Chemoradiotherapy Group: Participants will receive carboplatin (AUC=2) IV and paclitaxel (50mg/m²) IV on day 1,8,15,22,29. And radiotherapy will start on day 1 of chemotherapy. A total of 41.4 Gy, 23 fractions of 1.8 Gy, 5 fractions a week. Participants will also receive pembrolizumab (2mg/kg) IV on days 1 and 22. Surgery will be performed within 4-6 weeks after completion of preoperative therapy described above.
Period: Overall Study
Arm/Group | Preoperative Pembrolizumab With Chemoradiotherapy Group
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Preoperative Pembrolizumab With Chemoradiotherapy Group
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] | 62 [42 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 20
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 20
Body Mass Index (BMI) [Median (Full Range); unit: kg/m^2] | 23.20 [15.31 to 29.06]
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Brief description of the criteria of Eastern Cooperative Oncology Group (ECOG) Performance Status: grade 0, normal activity; grade 1, restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; grade 2, capable of all selfcare but unable to carry out any work activities, ambulatory for more than 50% of time; grade 3, ambulatory for less than 50% of time, capable of only limited selfcare; grade 4, completely disabled, can not carry on any selfcare, totally confined to bed or chair; grade 5, dead.
  Participants
    0 | 3
    1 | 17
Smoking History [Count of Participants; unit: Participants]
  Non-smoker | 6
  Previous or current smoker | 14
Tumor Length [Median (Full Range); unit: cm] | 6.34 [3.70 to 13.00]
Tumor Location [Count of Participants; unit: Participants]
  Proximal third | 5
  Middle third | 11
  Distal third | 4
Clinical T Stage [Count of Participants; unit: Participants] — Clinical T stage was measured according to the American Joint Committee on Cancer criteria for esophageal carcinoma, eighth edition, and was evaluated based on pretreatment examinations, including physical examination, contrast-enhanced chest computed tomography, PET-CT, upper gastrointestinal endoscopy, etc. cT3 refers to tumor which invades the adventitia. cT4a refers to tumor which invades the pleura, pericardium, azygos vein, diaphragm, or peritoneum.
  Participants
    cT3 | 16
    cT4a | 4
Clinical N Stage [Count of Participants; unit: Participants] — Clinical N stage was measured according to the American Joint Committee on Cancer criteria for esophageal carcinoma, eighth edition, and was evaluated based on pretreatment examinations, including physical examination, contrast-enhanced chest computed tomography, PET-CT, upper gastrointestinal endoscopy, etc. Brief description of the criteria: cN0, no regional lymph node metastasis; cN1, metastasis in 1-2 regional lymph nodes; cN2, metastasis in 3-6 regional lymph nodes; cN3, metastasis in ≥7 regional lymph nodes.
  Participants
    cN0 | 2
    cN1 | 5
    cN2 | 10
    cN3 | 3
Clinical Stage [Count of Participants; unit: Participants] — Clinical stage refers to cTNM stage, which was measured based on the American Joint Committee on Cancer criteria for esophageal carcinoma, eighth edition. cT2N0-1M0 and cT3N0M0 are grouped into stage II. cT1-3N2M0 and cT3N1 are grouped into stage III. cT4a-4bN0-3M0 and cT1-3N3 are grouped into stage IVA. As the clinical stage increases, the severity of the esophageal cancer increases.
  Participants
    II | 2
    III | 13
    IVA | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety (Number of Participants With Grade 3 and Higher-grade Treatment-related Adverse Events)
Description: The number of participants with grade 3 and higher-grade treatment-related adverse events. Adverse events were evaluated using CTCAE 4.0, grade 3 treatment-related adverse events and higher-grade adverse events were reported.
Time Frame: From date of treatment allocation until surgery was applied during study period or up to at least 90 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Pembrolizumab With Chemoradiotherapy Group
Number analyzed (Participants) | 20
Participants | 13

2. Secondary Outcome: Feasibility (Number of Participants Who Finished Pembrolizumab With Chemoradiotherapy and Receive Surgery Within 4-6 Weeks After Preoperative Therapies)
Description: The number of participants who finished pembrolizumab with chemoradiotherapy and receive surgery within 4-6 weeks after preoperative therapies.
Time Frame: From date of treatment allocation until surgery or definitive chemoradiotherapy was applied, whichever came first, assessed up to 5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Pembrolizumab With Chemoradiotherapy Group
Number analyzed (Participants) | 20
Participants | 11

3. Secondary Outcome: Pathologic Complete Response
Description: Pathologic complete response was defined as the lack of all signs of cancer in tissue samples removed during surgery after treatment with pembrolizumab and chemoradiotherapy.
Time Frame: Two weeks after surgery
Population: Twenty patients were assigned to this group, while, 18 patients received esophagectomy. Two patients did not receive surgery due to the following reasons: one was determined progression disease due to liver metastasis after completion of preoperative therapy; another patient died while awaiting surgery due to severe esophageal hemorrhage.
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Pembrolizumab With Chemoradiotherapy Group
Number analyzed (Participants) | 18
Participants | 10

4. Secondary Outcome: Radiographic Response
Description: To assess radiographic response to neoadjuvant pembrolizumab with concurrent chemoradiotherapy using RECIST 1.1. Complete metabolic response (cMR), defined as a physiological distribution of FDG uptake on PET-CT with a SUVmax value of less than 4 with no nodal uptake.
Time Frame: From date of treatment allocation and during treatment period up to 3 months
Population: Twenty patients were enrolled, and seventeen patients out of them received PET-CT before and after the completion of preoperative treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Preoperative Pembrolizumab With Chemoradiotherapy Group
Number analyzed (Participants) | 17
Participants | 6

ADVERSE EVENTS:
Time Frame: From date of treatment allocation until surgery was applied during study period or up to at least 90 days after last dose.
Description: Adverse events were evaluated using Common Terminology Criteria for Adverse Events (CTCAE) 4.0.
Arm/Group | Preoperative Pembrolizumab With Chemoradiotherapy Group
All-Cause Mortality (participants affected / at risk) | 1/20
Serious Adverse Events (participants affected / at risk) | 13/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Preoperative Pembrolizumab With Chemoradiotherapy Group (N=20)
Leukopenia (Blood and lymphatic system disorders) | 2 — Grade 3 and higher-grade adverse events based on CTCAE 4.0.
Decreased neutrophil count (Blood and lymphatic system disorders) | 1 — Grade 3 and higher-grade adverse events based on CTCAE 4.0.
Lymphopenia (Blood and lymphatic system disorders) | 12 — Grade 3 and higher-grade adverse events based on CTCAE 4.0.
Esophageal hemorrhage (Gastrointestinal disorders) | 1 — Grade 3 and higher-grade adverse events based on CTCAE 4.0.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Preoperative Pembrolizumab With Chemoradiotherapy Group (N=20)
Leukopenia (Blood and lymphatic system disorders) | 18 — Adverse events during neoadjuvant therapy.
Decreased neutrophil count (Blood and lymphatic system disorders) | 8 — Adverse events during neoadjuvant therapy.
Lymphopenia (Blood and lymphatic system disorders) | 8 — Adverse events during neoadjuvant therapy.
Anemia (Blood and lymphatic system disorders) | 16 — Adverse events during neoadjuvant therapy.
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 — Adverse events during neoadjuvant therapy.
Alopecia (General disorders) | 11 — Adverse events during neoadjuvant therapy.
Anorexia (General disorders) | 9 — Adverse events during neoadjuvant therapy.
Constipation (Gastrointestinal disorders) | 4 — Adverse events during neoadjuvant therapy.
Diarrhea (Gastrointestinal disorders) | 2 — Adverse events during neoadjuvant therapy.
Fatigue (General disorders) | 11 — Adverse events during neoadjuvant therapy.
Nausea (Gastrointestinal disorders) | 8 — Adverse events during neoadjuvant therapy.
Vomiting (Gastrointestinal disorders) | 3 — Adverse events during neoadjuvant therapy.
Esophagitis (Gastrointestinal disorders) | 11 — Adverse events during neoadjuvant therapy.
Postoperative Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Anastomotic leakage (Respiratory, thoracic and mediastinal disorders) | 1/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Gastrointestinal fistula (Gastrointestinal disorders) | 1/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Wound infection (Skin and subcutaneous tissue disorders) | 1/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Hoarseness (Injury, poisoning and procedural complications) | 4/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Dysphagia (Gastrointestinal disorders) | 1/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.
Postoperative intrathoracic hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1/18 — Postoperative adverse events, which were assessed for 18 participants who underwent surgery.

LIMITATIONS AND CAVEATS:
This was a single arm study. The sample size was small. Patients were highly selected and from a single center. These may strict the generalizability of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03792347/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03792347/ICF_001.pdf